CLINICAL TRIAL: NCT03577288
Title: Impact of Appearance and Control of Emotions in Virtual Reality on Behaviour in Children and Young Adults: Link With Feeling of Presence
Brief Title: Impact of Emotion in Virtual Reality on Behavior of Children and Young Adults
Acronym: EPREV-EA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study had to be stopped in 2020 with the health crisis linked to COVID-19. Following this, and in view of the sanitary conditions, it was not possible to resume recruitment (research was taking place within the University of Lyon 2 and in schools)
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 69HCL18_0224
Record Dates: First submitted 2018-06-22; First posted 2018-07-05 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Healthy Volunteers
Keywords: Feelings; Emotions; Virtual Reality; Young Adult; Child

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experiment 1 A, B - Level of realism of EVR (Experimental): Participants (50 children and 50 young adults for part A, and 50 other children and 50 other young adults) will be exposed to virtual experience having different level of realism. In one condition the realism will be high (very close to the real word) and in the second condition the realism will be low (comparable to cartoon). The stimuli of interest included in virtual experience will be of three emotional categories : negative, positive and neutral.
  Interventions: Behavioral: manipulation of the level of realism
- Experiment 2 - Presence and size of avatar (Experimental): Participants (50 children and 100 young adults) will be exposed to virtual experiences in which in one condition they will be part of the virtual environment in a body of an avatar and in another condition the avatar will not be present.
  Children will be exposed to only one of the two possible situations: with an avatar or without an avatar for the entire experience. Adults will be exposed to only one of the four possible situations: with standard size avatar, with giant avatar, with tiny avatar, or without avatar.
  Interventions: Behavioral: manipulation of the presence and size of avatar
- Experiment 3 - Interaction in virtual experience (Experimental): Participants (50 children and 50 young adults) will be submitted to two conditions of virtual experience, one condition in which it is possible to interact with the stimuli presented in the virtual environment and another condition in which it is not possible to interact. In addition, the stimuli of interest will be of one of three emotional categories : negative, positive and neutral. Thus participants will be exposed to six short virtual experiences.
  Interventions: Behavioral: manipulation of interaction
- Experiment 4 - Animate/Inanimate nature of interactive objects (Experimental): Participants (30 children and 30 young adults) will be exposed to the virtual experience during which they will be able to interact in one condition with animated (e.g., dog, bird) stimuli and in another condition with inanimate (e.g., book, jacket) stimuli. The animate and inanimate stimuli of interest will be of three emotional categories : negative, positive and neutral.
  Interventions: Behavioral: manipulation of the nature of stimulus

INTERVENTIONS:
Behavioral: manipulation of the level of realism — The realism of the virtual experience will be manipulated. In one condition the realism will be high and in another condition the realism will be low. In addition, emotional category of stimuli for each virtual experience condition will be manipulated. Thus, each participant will be submitted to six virtual experiences (e.g., high realism with negative stimuli, low realism with negative stimuli, high realism with positive stimuli).
  The measures of the pupillary responses, gaze fixation, heart rate, head movement (only in part A) and Late Positive Potential (EEG - only in part B) will be realized. In addition, the participants will respond to the scales and questionnaire evaluating their emotion, feeling of presence and feeling of immersion.
  Arms: Experiment 1 A, B - Level of realism of EVR
Behavioral: manipulation of the presence and size of avatar — The presence of avatar in the virtual experience will be manipulated. In one condition the avatar will be present and in another condition the avatar will not be present. In addition, emotional category of stimuli for each virtual experience condition will be manipulated. Thus, each participant will be submitted to six virtual experiences (e.g., with avatar and negative stimuli, without avatar and negative stimuli, with avatar and positive stimuli, etc.).
  Children will be exposed to only one of the two possible situations: with an avatar or without an avatar for the entire experience. Adults will be exposed to only one of the four possible situations: with standard size avatar, with giant avatar, with tiny avatar, or without avatar.
  The measures of the pupillary responses, gaze fixation, heart rate, head movement will be realized. In addition, the participants will respond to the scales and questionnaire evaluating their emotion, feeling of presence and feeling of immersion.
  Arms: Experiment 2 - Presence and size of avatar
Behavioral: manipulation of interaction — Virtual experience condition will be manipulated. In one condition the participants will be exposed to the virtual experience in which they will be able to interact with some of the stimuli, in another condition they will not be able to interact with the stimuli (passive watching). In addition, emotional category of stimuli for each virtual experience condition will be manipulated. Thus, each participant will be submitted to six virtual experiences (e.g., interaction possible - negative stimuli, interaction impossible - negative stimuli, interaction possible - positive stimuli).
  The measures of the pupillary responses, gaze fixation, heart rate, head movement will be realized. In addition, the participants will respond to the scales and questionnaire evaluating their emotion, feeling of presence and feeling of immersion.
  Arms: Experiment 3 - Interaction in virtual experience
Behavioral: manipulation of the nature of stimulus — The nature of the stimuli with which the participants will interact will be manipulated. During virtual experience the participants will have a choice to interact or not with the virtual environment, in one condition with animate stimuli and in another condition with inanimate stimuli. In addition, emotional category of animate and inanimate stimuli will be manipulated. Thus, each participant will be submitted to six virtual experiences (e.g., condition with animate negative stimuli, condition with inanimate negative stimuli, condition with animate positive stimuli). The measures of the pupillary responses, gaze fixation, heart rate, head movement will be realized. In addition, the participants will respond to the scales and questionnaire evaluating their emotion, feeling of presence and feeling of immersion.
  Arms: Experiment 4 - Animate/Inanimate nature of interactive objects

SUMMARY:
Recently, researchers in the field of cognitive psychology have shown a great interest in Virtual Reality (VR). Indeed, this technology is the most advanced to create immersion and sense of presence in a virtual environment (VE) and gives the opportunity to study cognitive mechanisms in more ecological way. However, little is known about the impact of VR on the cognition and emotional states of the VR users. According to the scientific literature, the sense of presence (the fact that the user experiences the sense of being in the VE) is strongly related to the emotional experience, but it is not clear what mechanisms underline this relation. Thus, more research is necessary to its better understanding. Moreover, a few studies have shown age related differences in sense of presence, with children having greater inclination for sense of presence than adults. This might be explained by the fact that frontal cortex (which is responsible for a control of the sense of presence) is still developing in childhood (the maturation last for the beginning of adulthood).

The goal of the present study is to examine which factors might be responsible of the interaction between the sense of presence, the immersion and the emotional experience in Virtual Reality, and the age-related difference. Thus, the investigator study 2 types of healthy participants (volunteers) in order to examine the age-related difference in this interaction: young adults between 18 and 25 years old and children between 8 to 14 years old. To study different factors potentially involved in the interaction four experiments will be conducted. In each experiment the investigator manipulate one type of factor to study its impact on emotions and the sense of presence in a VE: (1) the image quality, (2) the fact that participant had an avatar (body) in the VE, (3) the possibility to interact or not in VE and (4) the nature of elements with which it is possible to interact (objects or living being). In the end of this study the investigator hope to contribute to the knowledge of adapted use of VR for different type of users, such as children and young adults.

ELIGIBILITY:
Inclusion Criteria:

Children:

* Age comprised between 8 and 14
* Native French speaker
* Two parents gave their informed consent for a participation of their child in the study

Young adults :

* Students
* Age comprised between 18 and 25
* Native French speaker
* Participant gave his/her informed consent for a participation in the study
* Participant has health insurance

Exclusion Criteria:

Children:

* Neurodevelopmental deficits, diagnosis of intellectual deficiency (Scores below 70 for Vineland II scale et Total IQ Total below 70 for WPPSI-IV (Wechsler, 2014) or WISC-V (Wechsler, 2016)) new by parents or legal representative
* Learning disorder (difficulties in learning and using scholar skills since at least 6 months new by teacher, parents or legal representative)
* History of psychiatric disorder new by parents or legal representative
* Neurological disorders new by parents or legal representative
* Drugs intake having impact on motor, cognitive or memory capacities (e.g., corticoids) new by parents or legal representative
* Visual or hearing disorders without correction
* Epilepsy
* Child, parents or legal representative no agreement to participate to the study

Young Adults :

* Neurological disorders new by participants
* Drugs intake having impact on motor, cognitive or memory capacities (e.g., corticoids)
* History of psychiatric disorder new by participant
* Use of drugs of alcohol
* Visual or hearing disorders without correction
* Epilepsy
* No agreement to participate to the study

Ages: 8 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 240 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
measure of valence and arousal with Self-Assessment Manikin (SAM) scale | Day 0
  Evaluation of emotion
response to the presence questionnaire (PQ, Witmer & Singer, 1998 | Day 0
  Evaluation of feeling of presence questionnaire PQ, Witmer & Singer, 1998
evaluation of feeling of immersion by a Likert scale | Day 0
  Evaluation of feeling of immersion
responses evoked by the stimuli of interest | Day 0
  During Experience in Virtual Reality (EVR) we will measure responses evoked by the stimuli of interest: with oculometer time fixation and pupillary dilatation, and with oximeter heart rate
Measure of evoked potential | Day 0
  During EVR only in Experiment 1B we will measure, using EEG, evoked potential, particularly Late Positive Potential (LPP)
Measure of head movements evoked by the stimuli of interest | Day 0
  During EVR except Experiment 1B we will measure, using the device integrated in VR equipment, head movements evoked by the stimuli of interest

CONTACTS AND LOCATIONS:
Overall Officials: Hanna CHAINAY, Principal Investigator — Université Lyon 2
Locations (1):
- EA3082 Laboratoire d'Etude des Mécanismes Cognitifs Institut de Psychologie Université Lyon 2, Bron, France